CLINICAL TRIAL: NCT01210989
Title: A Randomized,Placebo-controlled,Double-blind Trial of Phyllanthus Urinaria (Hepaguard®) in Adults With Nonalcoholic Steatohepatitis
Brief Title: Trial of Hepaguard® in Adults With Nonalcoholic Steatohepatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Henry LY Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAFLD- Hepaguard
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hepaguard (Active Comparator)
  Interventions: Drug: Phyllanthus urinaria
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Phyllanthus urinaria — Subjects meeting the inclusion and exclusion criteria will be randomized (2:1) to receive oral Hepaguard 1 g three times daily or placebo of identical appearance. At week 24, subjects receiving active Hepaguard will be randomized (1:1) to continue Hepaguard for another 24 weeks or stop treatment.
  Other Names: Hepaguard®
  Arms: Hepaguard
Drug: Placebo — Subjects meeting the inclusion and exclusion criteria will be randomized (2:1) to receive oral Hepaguard 1 g three times daily or placebo of identical appearance.
  Arms: Placebo

SUMMARY:
Nonalcoholic fatty liver disease is one of the most common chronic liver diseases worldwide. Nonalcoholic steatohepatitis (NASH) is the active form of the disease which runs a progressive course and may result in liver cirrhosis and liver cancer. However, there is yet proven treatment for this disorder. In cell line and animal studies, we have shown that Phyllanthus urinaria can ameliorate NASH by reducing oxidative stress and lipid accumulation. Phyllanthus (Hepaguard) has been used widely by patients with chronic liver diseases, but the efficacy in NASH has not been confirmed in humans.

This study is divided into two parts. In part 1, 60 patients with histology-confirmed NASH will be randomized to receive Hepaguard or placebo for 24 weeks to test the efficacy. Endpoints will be assessed at week 24. The aim of part 2 is to test the durability of Hepaguard. Forty patients originally on Hepaguard will be randomized again to continue Hepaguard for another 24 weeks or stop the treatment. The endpoints at week 48 will be further analyzed.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the most common chronic liver disease in affluent countries. Patients with nonalcoholic steatohepatitis (NASH), a severe form of NAFLD characterized by ballooning, lobular inflammation and liver fibrosis, have increased mortality rate and risk of cardiovascular disease. Besides, some patients progress to cirrhosis and may even develop hepatocellular carcinoma. In long-term studies, up to 13% of NAFLD patients died of hepatic complications.(1)

Owing to westernization of lifestyle, NAFLD is also increasing dramatically in Asia. In a population screening study in Shanghai using ultrasonography, 15% of adult Chinese was found to suffer from NAFLD.(2) Among Chinese patients with NAFLD, significant necroinflammation and liver fibrosis are not uncommon.(3-5) These patients also often have progression of liver fibrosis with time.(6)

Since NASH is closely related to type 2 diabetes and obesity, a logical approach would be to improve these metabolic parameters.(7, 8) Observational studies suggest that regular exercise and weight reduction benefit NASH patients. At present, there is no registered drug for the treatment of NASH. Although insulin sensitizers such as pioglitazone and rosiglitazone may improve the metabolic profile and hepatic necroinflammation,(9, 10) the effects are not durable.(11) Weight gain and cardiovascular complications also limit the use of these agents.(12, 13) More effective and better tolerated treatment is urgently needed.

Phyllanthus urinaria (Hepaguard®) is commonly used by patients with various chronic liver diseases.(14-16) Phyllanthus has excellent safety profile. In in vitro and in vivo models of NAFLD, Phyllanthus reduces hepatic steatosis, necroinflammation and fibrosis.(16) Oxidative stress and lipid accumulation are ameliorated. Whether the same beneficial effects apply to humans is unclear.

References:

1. Adams LA, Lymp JF, St Sauver J, Sanderson SO, Lindor KD, Feldstein A, Angulo P. The natural history of nonalcoholic fatty liver disease: a population-based cohort study. Gastroenterology 2005;129:113-21.
2. Fan JG, Zhu J, Li XJ, Chen L, Li L, Dai F, Li F, Chen SY. Prevalence of and risk factors for fatty liver in a general population of Shanghai, China. J Hepatol 2005;43:508-14.
3. Wong VW, Chan HL, Hui AY, Chan KF, Liew CT, Chan FK, Sung JJ. Clinical and histological features of non-alcoholic fatty liver disease in Hong Kong Chinese. Aliment Pharmacol Ther 2004;20:45-9.
4. Wong VW, Wong GL, Chim AM, Tse AM, Tsang SW, Hui AY, Choi PC, Chan AW, So WY, Chan FK, Sung JJ, Chan HL. Validation of the NAFLD fibrosis score in a Chinese population with low prevalence of advanced fibrosis. Am J Gastroenterol 2008;103:1682-8.
5. Wong VW, Wong GL, Tsang SW, Hui AY, Chan AW, Choi PC, Chim AM, Chu S, Chan FK, Sung JJ, Chan HL. Metabolic and histological features of non-alcoholic fatty liver disease patients with different serum alanine aminotransferase levels. Aliment Pharmacol Ther 2009;29:387-96.
6. Hui AY, Wong VW, Chan HL, Liew CT, Chan JL, Chan FK, Sung JJ. Histological progression of non-alcoholic fatty liver disease in Chinese patients. Aliment Pharmacol Ther 2005;21:407-13.
7. Wong VW, Hui AY, Tsang SW, Chan JL, Tse AM, Chan KF, So WY, Cheng AY, Ng WF, Wong GL, Sung JJ, Chan HL. Metabolic and adipokine profile of Chinese patients with nonalcoholic fatty liver disease. Clin Gastroenterol Hepatol 2006;4:1154-61.
8. Wong VW, Hui AY, Tsang SW, Chan JL, Wong GL, Chan AW, So WY, Cheng AY, Tong PC, Chan FK, Sung JJ, Chan HL. Prevalence of undiagnosed diabetes and postchallenge hyperglycaemia in Chinese patients with non-alcoholic fatty liver disease. Aliment Pharmacol Ther 2006;24:1215-22.
9. Belfort R, Harrison SA, Brown K, Darland C, Finch J, Hardies J, Balas B, Gastaldelli A, Tio F, Pulcini J, Berria R, Ma JZ, Dwivedi S, Havranek R, Fincke C, DeFronzo R, Bannayan GA, Schenker S, Cusi K. A placebo-controlled trial of pioglitazone in subjects with nonalcoholic steatohepatitis. N Engl J Med 2006;355:2297-307.
10. Ratziu V, Giral P, Jacqueminet S, Charlotte F, Hartemann-Heurtier A, Serfaty L, Podevin P, Lacorte JM, Bernhardt C, Bruckert E, Grimaldi A, Poynard T. Rosiglitazone for nonalcoholic steatohepatitis: one-year results of the randomized placebo-controlled Fatty Liver Improvement with Rosiglitazone Therapy (FLIRT) Trial. Gastroenterology 2008;135:100-10.
11. Lutchman G, Modi A, Kleiner DE, Promrat K, Heller T, Ghany M, Borg B, Loomba R, Liang TJ, Premkumar A, Hoofnagle JH. The effects of discontinuing pioglitazone in patients with nonalcoholic steatohepatitis. Hepatology 2007;46:424-9.
12. Balas B, Belfort R, Harrison SA, Darland C, Finch J, Schenker S, Gastaldelli A, Cusi K. Pioglitazone treatment increases whole body fat but not total body water in patients with non-alcoholic steatohepatitis. J Hepatol 2007;47:565-70.
13. Juurlink DN, Gomes T, Lipscombe LL, Austin PC, Hux JE, Mamdani MM. Adverse cardiovascular events during treatment with pioglitazone and rosiglitazone: population based cohort study. BMJ 2009;339:b2942.
14. Wang M, Cheng H, Li Y, Meng L, Zhao G, Mai K. Herbs of the genus Phyllanthus in the treatment of chronic hepatitis B: observations with three preparations from different geographic sites. J Lab Clin Med 1995;126:350-2.
15. Chan HL, Sung JJ, Fong WF, Chim AM, Yung PP, Hui AY, Fung KP, Leung PC. Double-blinded placebo-controlled study of Phyllanthus urinaris for the treatment of chronic hepatitis B. Aliment Pharmacol Ther 2003;18:339-45.
16. Shen B, Yu J, Wang S, Chu ES, Wong VW, Zhou X, Lin G, Sung JJ, Chan HL. Phyllanthus urinaria ameliorates the severity of nutritional steatohepatitis both in vitro and in vivo. Hepatology 2008;47:473-83.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above,
* Histologic NAFLD activity score 3,
* Written informed consent

Exclusion Criteria:

* Positive hepatitis B surface antigen, or anti-hepatitis C virus antibody, or histologic features of an alternative liver disease,
* Alcohol consumption above 30g per week in men or 20g per week in women,
* Serum alanine aminotransferase above 10 times the upper limit of normal,
* Liver decompensation,
* Evidence of hepatocellular carcinoma currently or in the past 5 years,
* Type 1 diabetes or insulin treatment,
* Use of investigational drugs in the last 12 weeks,
* Terminal illness or cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Histologic NAFLD activity score | week 24

SECONDARY OUTCOMES:
ALT normalization | week 24 & week 48
Metabolic endpoints | Weeks 12, 24, 36 and 48
Changes in magnetic resonance spectroscopy | Weeks 24 and 48
Liver stiffness measurement | Weeks 24 and 48
Biomarkers of NASH and liver fibrosis | Weeks 12, 24, 36 and 48

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Suen Man Shook Hepatitis Center, Institute of Digestive Disease, The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong SAR, China

REFERENCES:
- [Background] Adams LA, Lymp JF, St Sauver J, Sanderson SO, Lindor KD, Feldstein A, Angulo P. The natural history of nonalcoholic fatty liver disease: a population-based cohort study. Gastroenterology. 2005 Jul;129(1):113-21. doi: 10.1053/j.gastro.2005.04.014. PMID 16012941
- [Background] Fan JG, Zhu J, Li XJ, Chen L, Li L, Dai F, Li F, Chen SY. Prevalence of and risk factors for fatty liver in a general population of Shanghai, China. J Hepatol. 2005 Sep;43(3):508-14. doi: 10.1016/j.jhep.2005.02.042. PMID 16006003
- [Background] Wong VW, Chan HL, Hui AY, Chan KF, Liew CT, Chan FK, Sung JJ. Clinical and histological features of non-alcoholic fatty liver disease in Hong Kong Chinese. Aliment Pharmacol Ther. 2004 Jul 1;20(1):45-9. doi: 10.1111/j.1365-2036.2004.02012.x. PMID 15225170
- [Background] Wong VW, Wong GL, Chim AM, Tse AM, Tsang SW, Hui AY, Choi PC, Chan AW, So WY, Chan FK, Sung JJ, Chan HL. Validation of the NAFLD fibrosis score in a Chinese population with low prevalence of advanced fibrosis. Am J Gastroenterol. 2008 Jul;103(7):1682-8. doi: 10.1111/j.1572-0241.2008.01933.x. Epub 2008 Jul 4. PMID 18616651
- [Background] Wong VW, Wong GL, Tsang SW, Hui AY, Chan AW, Choi PC, Chim AM, Chu S, Chan FK, Sung JJ, Chan HL. Metabolic and histological features of non-alcoholic fatty liver disease patients with different serum alanine aminotransferase levels. Aliment Pharmacol Ther. 2009 Feb 15;29(4):387-96. doi: 10.1111/j.1365-2036.2008.03896.x. Epub 2008 Nov 17. PMID 19035982
- [Background] Hui AY, Wong VW, Chan HL, Liew CT, Chan JL, Chan FK, Sung JJ. Histological progression of non-alcoholic fatty liver disease in Chinese patients. Aliment Pharmacol Ther. 2005 Feb 15;21(4):407-13. doi: 10.1111/j.1365-2036.2005.02334.x. PMID 15709991
- [Background] Wong VW, Hui AY, Tsang SW, Chan JL, Tse AM, Chan KF, So WY, Cheng AY, Ng WF, Wong GL, Sung JJ, Chan HL. Metabolic and adipokine profile of Chinese patients with nonalcoholic fatty liver disease. Clin Gastroenterol Hepatol. 2006 Sep;4(9):1154-61. doi: 10.1016/j.cgh.2006.06.011. Epub 2006 Aug 14. PMID 16904946
- [Background] Wong VW, Hui AY, Tsang SW, Chan JL, Wong GL, Chan AW, So WY, Cheng AY, Tong PC, Chan FK, Sung JJ, Chan HL. Prevalence of undiagnosed diabetes and postchallenge hyperglycaemia in Chinese patients with non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2006 Oct 15;24(8):1215-22. doi: 10.1111/j.1365-2036.2006.03112.x. PMID 17014580
- [Background] Belfort R, Harrison SA, Brown K, Darland C, Finch J, Hardies J, Balas B, Gastaldelli A, Tio F, Pulcini J, Berria R, Ma JZ, Dwivedi S, Havranek R, Fincke C, DeFronzo R, Bannayan GA, Schenker S, Cusi K. A placebo-controlled trial of pioglitazone in subjects with nonalcoholic steatohepatitis. N Engl J Med. 2006 Nov 30;355(22):2297-307. doi: 10.1056/NEJMoa060326. PMID 17135584
- [Background] Ratziu V, Giral P, Jacqueminet S, Charlotte F, Hartemann-Heurtier A, Serfaty L, Podevin P, Lacorte JM, Bernhardt C, Bruckert E, Grimaldi A, Poynard T; LIDO Study Group. Rosiglitazone for nonalcoholic steatohepatitis: one-year results of the randomized placebo-controlled Fatty Liver Improvement with Rosiglitazone Therapy (FLIRT) Trial. Gastroenterology. 2008 Jul;135(1):100-10. doi: 10.1053/j.gastro.2008.03.078. Epub 2008 Apr 8. PMID 18503774
- [Background] Lutchman G, Modi A, Kleiner DE, Promrat K, Heller T, Ghany M, Borg B, Loomba R, Liang TJ, Premkumar A, Hoofnagle JH. The effects of discontinuing pioglitazone in patients with nonalcoholic steatohepatitis. Hepatology. 2007 Aug;46(2):424-9. doi: 10.1002/hep.21661. PMID 17559148
- [Background] Juurlink DN, Gomes T, Lipscombe LL, Austin PC, Hux JE, Mamdani MM. Adverse cardiovascular events during treatment with pioglitazone and rosiglitazone: population based cohort study. BMJ. 2009 Aug 18;339:b2942. doi: 10.1136/bmj.b2942. PMID 19690342
- [Background] Wang M, Cheng H, Li Y, Meng L, Zhao G, Mai K. Herbs of the genus Phyllanthus in the treatment of chronic hepatitis B: observations with three preparations from different geographic sites. J Lab Clin Med. 1995 Oct;126(4):350-2. PMID 7561442
- [Background] Chan HL, Sung JJ, Fong WF, Chim AM, Yung PP, Hui AY, Fung KP, Leung PC. Double-blinded placebo-controlled study of Phyllanthus urinaris for the treatment of chronic hepatitis B. Aliment Pharmacol Ther. 2003 Aug 1;18(3):339-45. doi: 10.1046/j.1365-2036.2003.01671.x. PMID 12895219
- [Background] Shen B, Yu J, Wang S, Chu ES, Wong VW, Zhou X, Lin G, Sung JJ, Chan HL. Phyllanthus urinaria ameliorates the severity of nutritional steatohepatitis both in vitro and in vivo. Hepatology. 2008 Feb;47(2):473-83. doi: 10.1002/hep.22039. PMID 18157836
- [Background] Ekstedt M, Franzen LE, Mathiesen UL, Thorelius L, Holmqvist M, Bodemar G, Kechagias S. Long-term follow-up of patients with NAFLD and elevated liver enzymes. Hepatology. 2006 Oct;44(4):865-73. doi: 10.1002/hep.21327. PMID 17006923
- [Background] Kleiner DE, Brunt EM, Van Natta M, Behling C, Contos MJ, Cummings OW, Ferrell LD, Liu YC, Torbenson MS, Unalp-Arida A, Yeh M, McCullough AJ, Sanyal AJ; Nonalcoholic Steatohepatitis Clinical Research Network. Design and validation of a histological scoring system for nonalcoholic fatty liver disease. Hepatology. 2005 Jun;41(6):1313-21. doi: 10.1002/hep.20701. PMID 15915461
- [Background] Angulo P, Hui JM, Marchesini G, Bugianesi E, George J, Farrell GC, Enders F, Saksena S, Burt AD, Bida JP, Lindor K, Sanderson SO, Lenzi M, Adams LA, Kench J, Therneau TM, Day CP. The NAFLD fibrosis score: a noninvasive system that identifies liver fibrosis in patients with NAFLD. Hepatology. 2007 Apr;45(4):846-54. doi: 10.1002/hep.21496. PMID 17393509
- [Background] Sterling RK, Lissen E, Clumeck N, Sola R, Correa MC, Montaner J, S Sulkowski M, Torriani FJ, Dieterich DT, Thomas DL, Messinger D, Nelson M; APRICOT Clinical Investigators. Development of a simple noninvasive index to predict significant fibrosis in patients with HIV/HCV coinfection. Hepatology. 2006 Jun;43(6):1317-25. doi: 10.1002/hep.21178. PMID 16729309
- [Derived] Wong VW, Wong GL, Chan AW, Chu WC, Choi PC, Chim AM, Yiu KK, Yu J, Chan FK, Chan HL. Treatment of non-alcoholic steatohepatitis with Phyllanthus urinaria: a randomized trial. J Gastroenterol Hepatol. 2013 Jan;28(1):57-62. doi: 10.1111/j.1440-1746.2012.07286.x. PMID 23034128